CLINICAL TRIAL: NCT01521481
Title: Analgesic Efficacy of Ultrasound-guided Inguinal Field Block (Genitofemoral, Iliohypogastric and Ilioinguinal Nerve Block) for Inguinal Hernia Surgery.
Brief Title: Ultrasound-guided Inguinal Field Block (Genitofemoral, Iliohypogastric and Ilioinguinal Nerve Block) for Inguinal Hernia Surgery
Acronym: U-IFB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Ospedaliera San Gerardo di Monza (Other)
Responsible Party: Principal Investigator, Zhirajr Mokini M.D., Principal Investigator, Azienda Ospedaliera San Gerardo di Monza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AR HSG 03 2010
Record Dates: First submitted 2012-01-24; First posted 2012-01-30 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal | interventions — Anesthesia, Conduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Triple inguinal nerve block (Experimental): Ropivacaine 5 mg/ml
  Interventions: Other: Triple inguinal nerve block.
- Unilateral subarachnoid anesthesia (Active Comparator): Bupivacaine 10 mg/ml
  Interventions: Other: Unilateral subarachnoid anesthesia

INTERVENTIONS:
Other: Triple inguinal nerve block. — Ultrasound-guided genitofemoral, iliohypogastric and ilioinguinal nerve block with ropivacaine 5 mg/ml, 150 mg.
  Other Names: Regional anesthesia for the groin.
  Arms: Triple inguinal nerve block
Other: Unilateral subarachnoid anesthesia — Subarachnoid anesthesia with hyperbaric bupivacaine 10 mg/ml, 12 mg, homolateral to inguinal hernia.
  Other Names: Regional anesthesia for the groin.
  Arms: Unilateral subarachnoid anesthesia

SUMMARY:
The purpose of this study is to investigate the analgesic efficacy of an ultrasound-guided inguinal field block (block of the genitofemoral, iliohypogastric and ilioinguinal nerve).

DETAILED DESCRIPTION:
Inguinal hernia repair accounts for 10-15% of all operations in general surgery. Moderate to severe pain can occur at the first day after inguinal hernia repair in 25% of patients at rest and in 60% during activity. On day 6 after the operation the incidence can be as high as 11% at rest and 33% during activity.

Ultrasound imaging for regional anesthesia techniques have improved the success and safety rate of nerve blocks. We hypothesized that a procedure consisting of an ultrasound-guided inguinal field block (genitofemoral, iliohypogastric and ilioinguinal nerve block and incision line infiltration) could effectively control postoperative pain compared to selective unilateral subarachnoid anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* BMI (Body mass index) < 30
* Non severe liver, renal or cardiac disease
* No allergy or contraindications to any of the study drugs
* American Hernia Society Score type I-II-IV-V hernia
* No pain or chronic analgesic administration in the preoperative period
* No previous surgery of the inguinal region
* Normal coagulation parameters and platelet count (> 100.000).
* Dicumarol and aspirin suspension for > 7 days
* Correctly administrated premedication
* No systemic infections
* No contraindications to subarachnoid anesthesia

Exclusion Criteria:

* BMI (Body mass index) > 30
* Severe liver, renal or cardiac disease
* Allergy or contraindications to any of the study drugs
* American Hernia Society Score type III-VI-VII-0 hernia
* Pain or chronic analgesic administration in the preoperative period
* Previous surgery of the inguinal region
* Anormal coagulation parameters and platelet count (< 100.000).
* No dicumarol and aspirin suspension for > 7 days
* Incorrectly administrated premedication
* Systemic infections
* Contraindications to subarachnoid anesthesia

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2011-04; Primary Completion 2011-10 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Pain Intensity. | Up to 24 hours.
  Postoperative pain will be assessed by numeric ranking scale (numeric ranking scale NRS 0 to 10 points) at rest (static numeric ranking scale NRS) and during activity (dynamic numeric ranking scale NRS).

SECONDARY OUTCOMES:
Supplemental local anesthesia infiltration | During surgery, up to 2 hours.
  If needed, surgeons can infiltrate tissues with 15 ml of ropivacaine 5 mg/ml.
Conversion to general anesthesia. | During surgery, up to 2 hours
  Patients will receive remifentanil adjusted to maintain spontaneous breathing and conscious sedation with a Ramsay score = 2 during surgery if modest pain (numeric ranking scale NRS > 4 and agitation) is sustained. If remifentanil is not sufficient for restoring patient comfort, the block will be considered failed and the patient will be given general anesthesia with propofol and a Proseal Laryngeal Mask.
mPADSS (Post-Anesthesia Discharge Scoring System) | Up to 24 hours
  Assessed at every evaluation time postoperatively. The modified Post-Anesthesia Discharge Scoring System (mPADSS) includes stable heart and respiratory rates, absence of excessive nausea and pain, no bleeding from the surgical site, and ability to walk without support.
Analgesic requirement | Up to 7 days
  Assessed at every evaluation time postoperatively.
Activity | Up to 7 days
  Assessed through the activities assessment questionnaire 7 days after surgery.
Adverse events. | Up to 7 days
  Assessed at every evaluation time and including surgical and anesthesiological related events.
Time from the end of anesthesia to first micturition. | Up to 24 hours.
  Assessed at every evaluation time postoperatively.
Time from the end of surgery to the first unassisted walking. | Up to 24 hours.
  Assessed at every evaluation time postoperatively.
Total intrahospital stay. | Up to 24 hours.
  Assessed at every evaluation time postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Zhirajr Mokini, M.D., Principal Investigator — San Gerardo Hospital; Pablo Mauricio Ingelmo, M.D., Study Director — San Gerardo Hospital
Locations (1):
- San Gerardo Hospital, Monza, Italy